CLINICAL TRIAL: NCT00215098
Title: Chylothorax in Children Following Congenital Heart Surgery
Brief Title: Chylothorax Following Heart Surgery
Status: Terminated | Type: Observational
Why Stopped: insufficient data
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-093
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2007-06

CONDITIONS: Chylothorax
Keywords: pediatric health; cardiac; congenital heart surgery; post-operative chylous effusions; heart defects; children
MeSH Terms: conditions — Chylothorax

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine at risk populations for certain congenital heart defects or certain operative procedures and to define the associated morbidity secondary to chylothorax - prolonged chest tube drainage, prolonged hospital stay, need for central access and hyperalimentation, subsequent infection.

DETAILED DESCRIPTION:
Chylothorax is not uncommon following congenital heart surgery. It often results in prolonged chest tube drainage and hospital stays. Due to the feeding difficulties, it often results in malnutrition and the need for central hyperalimentation. In addition, it results in a depressed immune system with the possibility of subsequent infection. Chylothorax can be a significant contributor to post-operative morbidity and mortality.

The primary aims are to determine at risk populations - certain congenital heart defects or certain operative procedures, to define the associated morbidity secondary to chylothorax - prolonged chest tube drainage, prolonged hospital stay, need for central access and hyperalimentation, subsequent infection and to review our current treatment methods - change formulas, hyperalimentation, somatostatin. The secondary aims are to determine ways to prevent chylothorax, determine the most successful treatment method, and to discover better treatment methods. This study will be conducted through a retrospective chart review.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the congenital surgery database
* patients have developed post-operative chylous effusions

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the congenital surgery database
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2005-05; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kogon, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States